CLINICAL TRIAL: NCT00455689
Title: Understanding Experimentally Induced Hot Flushes and Their Impact on Sleep and Mood
Brief Title: Understanding Experimentally Induced Hot Flushes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Endocrine Research Society (Other)
Responsible Party: Principal Investigator, Hadine Joffe, MD, Vice Chair for Psychiatry Research, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2005P-001512
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Results first posted 2018-08-21 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-08

CONDITIONS: Hot Flashes
Keywords: Lupron; Premenopausal; Hot flashes
MeSH Terms: conditions — Hot Flashes | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Developed hot flashes (Experimental): Subjects who developed hot flashes after receiving leuprolide acetate (3.75 mg intramuscular injection)
  Interventions: Drug: Leuprolide acetate
- Did not develop hot flashes (Experimental): Subjects who did not develop hot flashes after receiving leuprolide acetate (3.75 mg intramuscular injection)
  Interventions: Drug: Leuprolide acetate

INTERVENTIONS:
Drug: Leuprolide acetate — Leuprolide acetate (Lupron Depot®) 3.75-mg intramuscular injection
  Leuprolide is a widely used gonadotropin-releasing hormone agonist (GnRHa) that is indicated for treatment of endometriosis, uterine fibroids, precocious puberty, and prostate cancer, and is used off-label for in-vitro fertilization and premenstrual syndrome. In this protocol, leuprolide will be administered once during the mid-luteal phase of the menstrual cycle at a dose routinely used for treatment of endometriosis and uterine fibroids in women.
  Other Names: Lupron

SUMMARY:
The purpose of the study is to examine the impact of hot flushes on sleep, mood, and well-being. The investigators will cause hot flushes by giving study participants the hormone medication, leuprolide (Lupron), which is a manufactured (artificial) hormone that makes the body think that it has reached menopause temporarily. Most women begin to have hot flushes within 4 weeks after taking leuprolide and resume menses 3 months later. The investigators will administer questionnaires to evaluate changes in sleep and mood over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-45 years old
* Premenopausal
* Willingness to use barrier methods of contraception during study and after completion of study until menses resume
* Good general health

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Hot flushes
* Hemoglobin at the screening visit less than 10 gm/dL
* Abnormal liver function tests
* Abnormal renal function tests
* BMI > 35 kg/m2
* Previously diagnosed osteoporosis or osteopenia
* Psychiatric disorder involving mood, anxiety, psychotic disorder, current anorexia nervosa, or current alcohol or substance-use disorder
* Previous severe depression
* Evidence of suicidal or homicidal ideation
* Sleep apnea, narcolepsy, or other diagnosed sleep disorder
* Contraindication, hypersensitivity, or previous allergic reaction to GnRH agonists
* Regular use of centrally active medications
* Use of hormonal medications for at least 2 months
* Use of ketoconazole, clomiphene citrate, or anabolic/androgenic steroids in the preceding 3 months
* Renal insufficiency
* Abnormal vaginal bleeding
* History of thrombo-embolism or cardiovascular disease
* History of congestive heart failure or other conditions requiring sodium restriction
* History of spinal cord compression
* Metastatic vertebral lesions
* Memory disorders
* Urinary tract obstruction
* History of liver, kidney, pulmonary, or metabolic disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-11-28 (Actual); Primary Completion 2007-07-24 (Actual); Study Completion 2007-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hadine Joffe, M.D., M.Sc., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Joffe H, Deckersbach T, Lin NU, Makris N, Skaar TC, Rauch SL, Dougherty DD, Hall JE. Metabolic activity in the insular cortex and hypothalamus predicts hot flashes: an FDG-PET study. J Clin Endocrinol Metab. 2012 Sep;97(9):3207-15. doi: 10.1210/jc.2012-1413. Epub 2012 Jun 20. PMID 22723326

RESULTS

PARTICIPANT FLOW:
Groups:
- Developed Hot Flashes: Subjects who developed hot flashes after receiving leuprolide acetate (3.75 mg intramuscular injection)
  Leuprolide acetate: Leuprolide acetate (Lupron Depot®) 3.75-mg intramuscular injection
  Leuprolide is a widely used GnRH agonist that is indicated for treatment of endometriosis, uterine fibroids, precocious puberty, and prostate cancer, and is used off-label for in-vitro fertilization and premenstrual syndrome. In this protocol, leuprolide will be administered once during the mid-luteal phase of the menstrual cycle at a dose routinely used for treatment of endometriosis and uterine fibroids in women.
- Did Not Develop Hot Flashes: Subjects who did not develop hot flashes after receiving leuprolide acetate (3.75 mg intramuscular injection)
  Leuprolide acetate: Leuprolide acetate (Lupron Depot®) 3.75-mg intramuscular injection
  Leuprolide is a widely used GnRH agonist that is indicated for treatment of endometriosis, uterine fibroids, precocious puberty, and prostate cancer, and is used off-label for in-vitro fertilization and premenstrual syndrome. In this protocol, leuprolide will be administered once during the mid-luteal phase of the menstrual cycle at a dose routinely used for treatment of endometriosis and uterine fibroids in women.
Period: Overall Study
Arm/Group | Developed Hot Flashes | Did Not Develop Hot Flashes
Started | 14 | 6
Completed | 14 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Developed Hot Flashes | Did Not Develop Hot Flashes | Total
Number analyzed (Participants) | 14 | 6 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (9.0) | 25.5 (6.7) | 30.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 20
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 8 | 3 | 11
  Hispanic or African-American | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Objective Sleep Efficiency
Description: Objective sleep efficiency was measured using actigraphy. Sleep efficiency (percent of time spent asleep between bedtime and wake time) was calculated and averaged over 2 consecutive nights both before and 4 weeks after receiving the intervention.
Time Frame: baseline (before receiving intervention) and 4 weeks after receiving intervention
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Developed Hot Flashes | Did Not Develop Hot Flashes
Number analyzed (Participants) | 14 | 6
percent change | -2.6 [-10.2 to -0.9] | 4.2 [0.8 to 7.5]

2. Secondary Outcome: Change in Subjective Sleep Quality
Description: Sleep quality was measured using the Pittsburgh Sleep Quality Index (PSQI; range 0-21, higher score indicates poorer quality sleep), which was administered both before and four weeks after receiving the intervention.
Time Frame: baseline (before receiving intervention) and 4 weeks after receiving intervention
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Developed Hot Flashes | Did Not Develop Hot Flashes
Number analyzed (Participants) | 14 | 6
units on a scale | 2.5 [1.0 to 4.0] | 1.0 [1.0 to 2.0]

ADVERSE EVENTS:
Time Frame: Subjects were monitored for 3 months following GnRHa administration
Groups:
- All Subjects: 20 subjects who all received one leuprolide injection
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 13/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=20)
Headache (Nervous system disorders) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
malodorous urine (Renal and urinary disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Irritability (Psychiatric disorders) | 1 (1)
Increased libido (General disorders) | 1 (1)
Edema (Vascular disorders) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes